CLINICAL TRIAL: NCT03737877
Title: The Feasibility of a Microbiome Dietary Intervention in Children With ADHD
Brief Title: The Feasibility of a Dietary Intervention in Children With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St Mary's University College (Other)
Collaborators: Goldsmiths, University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SMEC_2017-18_132
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: ADHD; Diet Modification
Keywords: ADHD; Diet Modification
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet modification (Experimental)
  Interventions: Other: Diet modification

INTERVENTIONS:
Other: Diet modification — The parents will have four group sessions with a nutritional therapist, where in depth advice and information about the diet will be provided. Ongoing support will also be provided throughout the study by use of a closed Facebook or WhatsApp group (whichever the parents choose as most appropriate). The diet is based on five main principles:
  * Eat at least seven portions of different varieties of fruit and vegetables each day.
  * Have a 12 hour overnight break from food (water only during this time).
  * Drink a Kefir drink each day - provided free of charge.
  * Eat a microbiome friendly, protein rich, breakfast from our menu.
  * Reduce sugar and artificial sweeteners.

SUMMARY:
The aim is to conduct a feasibility pilot study of a dietary intervention designed to optimise gut bacteria in children diagnosed with ADHD.

DETAILED DESCRIPTION:
Children with Attention Deficit Hyperactivity Disorder (ADHD) can suffer debilitating symptoms, including problematic behaviour and sleep. Research suggests dietary manipulations may be a helpful treatment option for children with ADHD, although the most effective are highly restrictive, with little known about why they might work. Optimising gut bacteria in individuals with ADHD may help alleviate some of the symptoms of this condition via the gut-brain-axis and would provide a plausible mechanism by which dietary interventions operate. We propose to conduct a feasibility pilot study of a dietary intervention designed to optimise gut bacteria in children diagnosed with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Parent-reported diagnosis of ADHD.
2. Children aged between 8 years - 13 years 11 months at onset of study.
3. Children not taking ADHD medication (such as methylphenidate) at the time of the study.
4. Parental permission to attend three group sessions and for themselves and their child to complete the requisite assessments.
5. Both males and females are eligible to take part.
6. Children with a co-occurring diagnosis will be accepted onto the trial.
7. Children with food allergies/sensitivities/coeliac disease will be accepted onto the trial.

Exclusion Criteria:

1. Children undergoing a current course of behavioural therapy.
2. Children currently on ADHD medication (such as methylphenidate).
3. Children who have taken antibiotics in the past 3 months

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Completion of study | final week
  What proportion of participants completed the study?

SECONDARY OUTCOMES:
Adherence to diet | week 6 of diet
  Percentage adherence to diet over the 4-week period based on parental report (range 0-100 % - high score reflecting greater degree of adherence).
Side-effects | duration of the 6 week diet
  Parent-reported side effects during course of study. (Qualitative) (More/more side-effects reflect poorer outcome).
The Conners Clinical Index (Conners CI) - Parent-report | Baseline and week 6 of diet
  Parental report of clinical symptoms (percentile score - higher score reflects more/more severe symptoms)
  1. Disruptive Behavior Indicator
  2. Learning and Language Disorder Indicator
  3. Mood Disorder Indicator
  4. Anxiety Disorder Indicator
  5. ADHD Indicator
The Conners Clinical Index (Conners CI) - Teacher-report | Baseline and week 6 of diet
  Teacher report of clinical symptoms (percentile score - higher score reflects more/more severe symptoms)
  1. Disruptive Behavior Indicator
  2. Learning and Language Disorder Indicator
  3. Mood Disorder Indicator
  4. Anxiety Disorder Indicator
  5. ADHD Indicator
The Conners Clinical Index (Conners CI) - Self-report | Baseline and week 6 of diet
  Child self-report of clinical symptoms (percentile score - higher score reflects more/more severe symptoms)
  1. Disruptive Behavior Indicator
  2. Learning and Language Disorder Indicator
  3. Mood Disorder Indicator
  4. Anxiety Disorder Indicator
  5. ADHD Indicator
Delayed Match to Sample test (Cambridge Neuropsychological Test Automated Battery - CANTAB) Latency (response time) Accuracy (correct patterns selected). | Baseline and week 6 of diet
  Computerised test of visual working memory
  * DMS Percent Correct (overall, for all delays, simultaneous, 0 sec delay, 4 sec delay, 12 sec delay). Range 0-100% - higher score reflects greater accuracy.
  * DMS Mean & Median Correct Latency (overall, for all delays, simultaneous, 0 sec delay, 4 sec delay, 12 sec delay). Range 0-∞ ms - higher score reflects worse performance.
  * DMS Correct Latency Standard Deviation. Range 0-∞ ms - higher score reflects worse performance.
  * DMS Mean Choices to Correct response. Range 0-4 - higher score reflects worse performance.
  * DMS Probability of Error Given Error. Range 0-1 - higher score reflects worse performance.
The Consensus Sleep Diary | Baseline and week 6 of diet
  Record of sleep - used qualitatively to detect and remove artefacts from the data.
Children's Sleep Habits Questionnaire | Baseline and week 6 of diet
  Parental report of child's sleep A Total Sleep Disturbances score is calculated as the sum of all CSHQ scored questions, and can range from 33 to 99. A higher score indicates more problematic sleep.
Sleep self-report questionnaire | Baseline and week 6 of diet
  Week long retrospective sleep survey (Scores range from 13-39 with a higher score indicating more/more severe sleep difficulties).
Actigraphy recordings | Baseline and week 6 of diet
  Objective measure of sleep quality and daytime activity
  * Mean activity during sleep. Range 0-∞. A higher score = less sound sleep (worse).
  * Minutes spent awake during the down period. Range 0-∞. A higher score = less sound sleep (worse).
  * Sleep latency (time taken to fall asleep). Range 0-∞. A higher score = more time taken to fall asleep (worse).
  * Sleep efficiency (% down period spent asleep, after removing sleep latency). A higher score = better.
  * Wake after sleep onset (minutes spent awake during the down period after removing sleep latency). Range 0-∞. A higher score = less sound sleep (worse).
  * Sleep fragmentation (number of awakenings/ total minutes of sleep x 100) - Higher score = more fragmented sleep (worse).
  * Mean daytime activity (0-∞) not necessarily worse or better.
The Gastrointestinal Symptom Rating | Baseline and week 6 of diet
  Questionnaire to evaluate common gastrointestinal symptoms Total scores range from 15-105 (with higher scores reflecting more/more severe gastrointestinal symptoms).
  Subscales:
  1. Abdominal pain (abdominal pain, hunger pains and nausea). Range 3-21 - a high score reflects worse symptoms.
  2. Reflux syndrome (heartburn and acid regurgitation). Range 3-21 - a high score reflects worse symptoms.
  3. Diarrhoea syndrome (diarrhoea, loose stools and urgent need for defecation). Range 3-21 - a high score reflects worse symptoms.
  4. Indigestion syndrome (borborygmus, abdominal distension, eructation and increased flatus). Range 3-21 - a high score reflects worse symptoms. Range 3-21 - a high score reflects worse symptoms.
  5. Constipation syndrome (constipation, hard stools and feeling of incomplete evacuation). Range 3-21 - a high score reflects worse symptoms.
Stool sample analysis for commensal bacteria and microbial diversity using 16S rRNA sequencing | Baseline and week 6 of diet
  Analysis of bacterial strains and diversity within stool sample
Treatment Acceptability Scale | Baseline and week 6 of diet
  Questionnaire to assess the acceptability of the diet to parents of the children taking part in the study Score range 6-42 (High score reflects more positive attitude to treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
At the request of individual researchers.

REFERENCES:
- [Derived] Lawrence K, Myrissa K, Toribio-Mateas M, Minini L, Gregory AM. Trialling a microbiome-targeted dietary intervention in children with ADHD-the rationale and a non-randomised feasibility study. Pilot Feasibility Stud. 2022 May 23;8(1):108. doi: 10.1186/s40814-022-01058-4. PMID 35606889